CLINICAL TRIAL: NCT02448680
Title: A Phase III Study on the Safety, Pharmacokinetics, and Efficacy of Coagulation Factor VIIa (Recombinant) in Congenital Hemophilia A or B Pediatric Patients From Birth to <12 Years Old With Inhibitors to Factor VIII or IX: PerSept 2
Brief Title: A Phase III Study on the Safety, Pharmacokinetics and Efficacy of Coagulation Factor VIIa
Acronym: PERSEPT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Collaborators: LFB USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LFB-FVIIa-007-14
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Hemophilia A With Inhibitors; Hemophilia B With Inhibitors
MeSH Terms: interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coagulation Factor VIIa (Recombinant): 75 µg/kg (Active Comparator): 75 µg/kg treatment regimen for 3 months
  Interventions: Biological: Coagulation FVIIa (Recombinant)
- Coagulation Factor VIIa (Recombinant): 225 µg/kg (Active Comparator): 225 µg/kg treatment regimen for 3 months
  Interventions: Biological: Coagulation FVIIa (Recombinant)

INTERVENTIONS:
Biological: Coagulation FVIIa (Recombinant) — A cross over design to assess the efficacy of 2 separate dose regimens (75 µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII or Factor IX

SUMMARY:
The purpose of the study is to assess the safety, efficacy and pharmacokinetics of 2 separate dose regimens (75µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII or IX in 12 patients ( birth to <6 years old), and 12 patients (≥6 years old to <12 years old).

DETAILED DESCRIPTION:
A Phase III Study on the Safety, Pharmacokinetics, and Efficacy of Coagulation Factor VIIa (Recombinant) in Congenital Hemophilia A or B Pediatric Patients from birth to <12 years old with Inhibitors to Factor VIII or IX: PerSept 2

ELIGIBILITY:
Inclusion Criteria:

* be male with a diagnosis of congenital hemophilia A or B of any severity
* have one of the following:
* a positive inhibitor test BU ≥5, OR
* a Bethesda Unit (BU) <5 but expected to have a high anamnestic response to FVIII or FIX, as demonstrated from the patient's medical history, precluding the use of factor VIII or IX products to treat bleeding episodes, OR
* a BU <5 but expected to be refractory to increased dosing of FVIII or FIX, as demonstrated from the patient's medical history, precluding the use of factor VIII or IX products to treat bleeding episodes
* be aged from birth to <12 years old
* have experienced at least 3 bleeding episodes of any severity in the past 6 months
* parents or legal guardians must be capable of understanding and be willing to comply with the conditions of the protocol
* parents or legal guardians must have read, understood, and provided written informed consent

Exclusion Criteria:

* have any coagulation disorder other than hemophilia A or B
* be immunosuppressed (i.e., the patient may not be receiving systemic immunosuppressive medication; cluster of differentiation 4 (CD4) counts at screening must be >200/µL)
* have a known allergy or hypersensitivity to rabbits
* have platelet count <100,000/mL
* have had a major surgical procedure (e.g. orthopedic, abdominal) within 1 month prior to first administration of study drug
* have received an investigational drug within 30 days of first study drug administration, or be expected to receive such drug during participation in this study

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, MD, Principal Investigator — University of Colorado, Denver
Locations (9):
- United States (3):
  - University of Colorado Denver Hemophilia & Thrombosis Center, Aurora, Colorado
  - Jimmy Everest Center for Cancer and Bleeding Disorders, Oklahoma City, Oklahoma
  - UT Southwestern Medical Center at Dallas / Children's Medical Center, Dallas, Texas
- University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Bulgaria
- University Hospital Motol, Prague, Czechia
- Hematology of Department Hemophilia and Thromboses center, Tbilisi, Georgia
- Worthwhile Clinical Trials, Benoni, South Africa
- Ukraine (2):
  - National Specialized Children's Hospital OKHMATDYT, Centre for Hemostatic Pathology (Ukraine), Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young G, Mahlangu J, Boggio LN, Carcao M, Dargaud Y, Escobar M, Giermasz A, Hermans C, Kuriakose P, Miesbach W, Nance D, Rafique A, Sidonio RF Jr, Vilchevska KV, Wang M, Pipe SW. Treatment of severe bleeds with eptacog beta in hemophilia A or B with inhibitors: a post hoc analysis of the PERSEPT 1 and 2 trials. Blood Vessel Thromb Hemost. 2025 Mar 27;2(3):100069. doi: 10.1016/j.bvth.2025.100069. eCollection 2025 Aug. PMID 40765904
- [Derived] Carcao M, Hermans C, Giermasz A, Kessler C, Miesbach W, Quon D, Windyga J, Mahlangu J. Safety and Use of Eptacog Beta 225 microg/kg in Patients With Haemophilia A or B With Inhibitors. Haemophilia. 2025 Sep;31(5):957-965. doi: 10.1111/hae.70083. Epub 2025 Jul 17. PMID 40674256

RESULTS

PARTICIPANT FLOW:
Groups:
- FVIIa: 75 µg/kg First, Then 225 µg/kg; FVIIa: 225 µg/kg First, Then 75 µg/kg: Coagulation Factor VIIa (Recombinant) : First Intervention (3 months), Second Intervention (3 months), repeat sequence for entirety of study.
Period: Overall Study
Arm/Group | FVIIa: 75 µg/kg First, Then 225 µg/kg | FVIIa: 225 µg/kg First, Then 75 µg/kg
Started | 12 | 13
Completed | 11 | 10
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FVIIa: 75 µg/kg First, Then 225 µg/kg | FVIIa: 225 µg/kg First, Then 75 µg/kg | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (3.02) | 4.8 (3.63) | 4.9 (3.28)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: Birth to < 6 years old | 6 | 7 | 13
  Age, Categorical: >= 6 years to < 12 years old | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 19.73 (7.432) | 21.94 (13.391) | 20.88 (10.782)
Height [Mean (Standard Deviation); unit: cm] | 104.21 (21.210) | 108.60 (25.904) | 106.49 (23.382)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 17.74 (2.505) | 17.35 (3.842) | 17.53 (3.209)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successfully Treated Mild/Moderate Bleeding Episodes Per FDA Requirement.
Description: For the primary efficacy endpoint, successful treatment of mild/moderate bleeding episode was defined as meeting all of the following:
  * "Good" or "excellent" response noted by the patient/parent/legal guardian or other caregiver, depending on patient's age and maturity
  * Study drug treatment: No further treatment with LR769 beyond timepoint where a "good" or "excellent" response for this bleeding episode was noted
  * No other hemostatic treatment needed for this bleeding episode
  * No administration of blood products that would indicate continuation of bleeding beyond timepoint where a "good" or "excellent" response for this bleeding episode was noted
  * No increase of pain beyond timepoint where a "good" or "excellent" response for this bleeding episode was noted that could not be explained other than as continuation of bleeding
Time Frame: 12 hours after first administration of study drug
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Proportion of successfully treated BEs
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- FVIIa 75 µg/kg: 75 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
- FVIIa 225µg/kg: 225 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes (BEs)) | 239 | 307
Proportion of successfully treated BEs | 0.654 [0.523 to 0.785] | 0.603 [0.482 to 0.723]

2. Primary Outcome: Proportion of Successfully Treated Bleeding Episodes (Mild/Moderate/Severe) Per EMA Definition
Description: * "Good" or "excellent" response noted by the patient/caregiver for mild/moderate bleeding episodes;
  * "Good" or "excellent" response noted by the physician for severe bleeding episodes.
Time Frame: 12 hours after first administration of study drug
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Proportion of successfully treated BEs
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- FVIIa 75 µg/kg: 75 µg/kg Treatment Regimen at Time of Bleeding Episode
- FVIIa 225 µg/kg: 225 µg/kg Treatment Regimen at Time of Bleeding Episode
Arm/Group | FVIIa 75 µg/kg | FVIIa 225 µg/kg
Number analyzed (Participants) | 23 | 24
Number analyzed (Bleeding Episodes (BEs)) | 239 | 310
Proportion of successfully treated BEs | 0.667 [0.533 to 0.800] | 0.625 [0.500 to 0.750]

3. Secondary Outcome: Patient-Reported "Good" or "Excellent" Response for Mild/Moderate Bleeding Episodes
Description: Based on Patient-Reported "Good" or "Excellent" responses as per the below descriptions:
  Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) had largely been reduced by the treatment, but had not completely disappeared. Symptoms had improved enough to not require more infusions of the study drug.
  Excellent: Full relief of pain and cessation of objective signs of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage). No additional infusion of study drug was required.
Time Frame: 12 hour after first administration of study drug
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Proportion of successfully treated BEs
Units Other Than Participants: Bleeding Episodes (BEs)
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes (BEs)) | 239 | 307
Proportion of successfully treated BEs | 0.667 [0.533 to 0.800] | 0.629 [0.502 to 0.756]

4. Secondary Outcome: Time to Patient Assessment of a "Good" or "Excellent" Response for Mild/Moderate Bleeding Episodes
Description: Categories of Response to Treatment are Described as Follows:
  None: No noticeable effect of the treatment on the bleed or worsening of patient's condition. Continuation of treatment with the study drug was needed.
  Moderate: Some effect of the treatment on the bleed was noticed, e.g., pain decreased or bleeding signs improved, but bleed continued and required continued treatment with the study drug.
  Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had largely been reduced by the treatment, but had not completely disappeared. Symptoms had improved enough to not require more infusions of the study drug.
  Excellent: Full relief of pain and cessation of objective signs of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage). No additional infusion of study drug was required.
Time Frame: Within 24 hours of Bleeding Episode
Population: Treated Population with non-missing measurements
Measure: Median (95% Confidence Interval); unit: Hours
Units Other Than Participants: Bleeding Episodes with Event
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes with Event) | 233 | 299
Hours | 9.00 [8.92 to 11.83] | 12.00 [11.83 to 12.00]

5. Secondary Outcome: Number of Administrations of Study Drug Per Mild/Moderate Bleeding Episode
Description: The number of study drug administrations with non-missing dose information in order to treat one mild/moderate bleeding episode.
Time Frame: Within 24 hours of Bleeding Episode
Population: Treated Population
Measure: Mean (Standard Deviation); unit: Administrations of Study Drug
Units Other Than Participants: Bleeding Episodes (BEs)
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes (BEs)) | 239 | 307
Administrations of Study Drug | 3.6 (2.27) | 2.6 (2.48)

6. Secondary Outcome: Total Amount of Study Drug Administered Per Mild/Moderate Bleeding Episode
Description: The total amount of study drug administered in order to treat one mild/moderate bleeding episode.
Time Frame: Within 24 hours of Bleeding Episode
Population: Treated Population with non-missing measurements
Measure: Mean (Standard Deviation); unit: mL per bleeding episode
Units Other Than Participants: Bleeding Episodes (BEs)
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes (BEs)) | 239 | 307
mL per bleeding episode | 6.733 (6.3693) | 8.287 (5.6531)

7. Other Pre Specified Outcome: Mild/Moderate Bleeding Episodes With Successful Pain Relief
Description: Successful pain relief was defined as a Visual Analogue Scale (VAS: 0-100; 0: no pain at all; 100: the worst pain ever possible) pain score at 12 hours after initial study drug administration that was less than the pain score at the start of treatment with study drug.
Time Frame: 12 hour after first administration of study drug
Population: Treated Population
Measure: Count of Units; unit: Bleeding Episodes (BEs)
Units Other Than Participants: Bleeding Episodes (BEs)
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 23 | 23
Number analyzed (Bleeding Episodes (BEs)) | 239 | 307
Bleeding Episodes (BEs) | 220 | 275

ADVERSE EVENTS:
Time Frame: From signing of the informed consent/assent until resolution or 30 days after the last dose of LR769 or early termination, whichever came first. The average duration for monitoring adverse event is about 11.2 months per patient.
Arm/Group | Coagulation Factor VIIa (Recombinant): 75 µg/kg | Coagulation Factor VIIa (Recombinant): 225 µg/kg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/25
Other Adverse Events (participants affected / at risk) | 12/23 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coagulation Factor VIIa (Recombinant): 75 µg/kg (N=23) | Coagulation Factor VIIa (Recombinant): 225 µg/kg (N=25)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) — Term from vocabulary, MedDRA 15.1
Paresis (Nervous system disorders) | 0 (0) | 1 (1) — Term from vocabulary, MedDRA 15.1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coagulation Factor VIIa (Recombinant): 75 µg/kg (N=23) | Coagulation Factor VIIa (Recombinant): 225 µg/kg (N=25)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Term from vocabulary, MedDRA 15.1
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) — Term from vocabulary, MedDRA 15.1
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) — Term from vocabulary, MedDRA 15.1
Bronchitis (Infections and infestations) | 1 (1) | 3 (4) — Term from vocabulary, MedDRA 15.1
Nasopharyngitis (Infections and infestations) | 4 (6) | 3 (3) — Term from vocabulary, MedDRA 15.1
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 2 (3) — Term from vocabulary, MedDRA 15.1
Rhinitis (Infections and infestations) | 3 (3) | 3 (3) — Term from vocabulary, MedDRA 15.1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) — Term from vocabulary, MedDRA 15.1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT02448680/Prot_001.pdf
  • Statistical Analysis Plan: Final Version 2.0 (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02448680/SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (v2.0) Addendum (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02448680/SAP_002.pdf